CLINICAL TRIAL: NCT04743401
Title: Feasibility of a Tele-game-based Exercise (Tele-exergame) Program to Prevent Deconditioning in Hospitalized COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: F3731-P; 42402 (Other: Baylor IRB)
Record Dates: First submitted 2021-01-12; First posted 2021-02-08 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: COVID 19; Rehabilitation; Inpatient; Hospitalized
Keywords: gaming; exer-gaming; telemedicine; inpatient; deconditioning; mobility; rehabilitation; virtual; persons under investigation for COVID; PUI
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: COVID-19 patients or PUI (persons under investigation) admitted to the MEDVAMC (n=60), with an anticipated length of stay of at least 3 days will be recruited. Participants will be randomized (n=1:1) to either intervention (IG) or control (CG) groups. Both groups will receive standard of care. IG will additionally receive Tele-Exergame MP therapy. Tele-Exergame sessions will range from 3-10 minutes based on patient ability and completed twice daily. They will complete assessments at baseline and at one-month post-hospital discharge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tele-exergame arm (Experimental): COVID-19 patients or PUI (persons under investigation) or other inpatients admitted to the MEDVAMC (n=60), with an anticipated length of stay of at least 3 days will be recruited. Participants will be randomized (n=1:1) to either intervention (IG) or control (CG) groups. Both groups will receive standard of care. IG will additionally receive Tele-Exergame MP therapy. Tele-Exergame sessions will range from 3-10 minutes based on patient ability and completed twice daily. They will complete assessments at baseline and at one-month post-hospital discharge.
  Interventions: Other: Tele-exergaming Tablet
- Convention care or control group (No Intervention): Standard of care only

INTERVENTIONS:
Other: Tele-exergaming Tablet — The Tele-Exergame platform virtually supervises exercise tasks and coaches patients to perform evidence-based foot and ankle exercises that have been designed to improve balance, cognition, and lower extremity vascular health.
  The exergame program uses a game-based approach, similar to playing a video game, which helps to increase patient motivation and engagement in the cognitively demanding exercise program.
  Arms: Tele-exergame arm

SUMMARY:
Background: Conventional face-to-face in-hospital mobility program (MP) is challenging for COVID-19 patients because of its associated risk of infection to hospital staff, staffing shortages as well as indirect risk of exposure to other hospitalized patients. Exergames are digital or web-based games that use body movement to promote physical activity and generally involve strength, balance, and flexibility exercises. The tele-exergame MP, developed by the team, uses a remotely supervised and game-based approach, which helps to increase patient motivation and engagement in a cognitively demanding exercise program.

Objectives: To demonstrate the feasibility, acceptability, and effectiveness of the Tele-Exergame mobility program in COVID-19 or PUI (persons under investigation), during hospitalization and examine post-hospitalization outcomes.

Research Design: Prospective randomized

DETAILED DESCRIPTION:
KEY RESEARCH AIMS:

Aim 1: To examine feasibility of Tele-exergame. The investigators will evaluate feasibility by documenting missing exercise sessions, exercise dropout, and acceptability questionnaire.

Aim 2: To examine proof of concept effectiveness to reduce deconditioning. The investigators will assess deconditioning (using wearables) and patient reported mental health assessed at baseline at discharge.

Aim 3: Examine proof of concept effectiveness to accelerate recovery post hospital discharge.

Approximately 4 weeks after discharge, patients will be contacted by telemedicine or telephone and requested to self-report on the Veterans mental health and the Veterans mobility.

METHODS:

COVID-19 patients or PUI (persons under investigation) admitted to the MEDVAMC (n=60), with an anticipated length of stay of at least 3 days will be recruited. Participants will be randomized (n=1:1) to either intervention (IG) or control (CG) groups. Both groups will receive standard of care. IG will additionally receive Tele-Exergame MP therapy. Tele-Exergame sessions will range from 3-10 minutes based on patient ability and completed twice daily. They will complete assessments at baseline and at one-month post-hospital discharge.

SCIENTIFIC MERIT:

The proposed contact-less mobility program could address the limitations of conventional in-hospital mobility program and advance the field of in-hospital exercise program.

The investigators will use innovative wearables to exploring potential digital biomarkers of hospital-acquired illness including cognitive-frailty. illness.

This study will advance the field of remote patient monitoring

BENEFIT TO VETERANS:

Its implementation not only for mobility program for hospitalized COVID-19 Veteran patients but also to deliver personalized exercise for non-COVID-19 Veteran patients with limited mobility including in bedbound and hospitalized Veteran patients Mobilizing hospitalized Veteran patients could mitigate hospital acquired complications like deconditioning, VTE and nosocomial infections and accelerate recovery post hospitalization

ELIGIBILITY:
Inclusion Criteria:

* Participants: Men or women Veterans with COVID-19 or PUI or hospitalized patients with duration of admission anticipated to be greater than 72 hours admitted to MEDVAMC.
* Length of stay: Anticipated length of stay at least 3 days.
* Ambulatory. Self-report of being ambulatory with or without an assistive device in the 2 weeks before admission.

Exclusion Criteria:

* ICU admission: The investigators will exclude those admitted to ICU at any point in their hospital stay.
* Admission of observation only: These patients will be excluded as length of stay is usually anticipated to be less than 3 days
* Median life expectancy: Those with imminently terminal (death expected in the next 30 days) will be excluded.
* Cognitive impairment: The investigators will exclude those with delirium, dementia, or severe cognitive impairment
* Medical condition: The investigators will exclude those who have any medical diagnosis deemed by the primary physician to be a contraindication to ambulation (i.e.: unstable from pulmonary embolus, unstable angina, severe hemodynamic instability etc.)
* Foot problem: The investigators will exclude those who have active foot ulcer or infection or major lower extremities amputation.
* Vision or hearing problems: The investigators will exclude those with hearing or visual problems that cannot be corrected with medical devices (glasses or hearing aids). Hearing or visual problems can limit their ability to interact with the exergame platform.
* lack of capacity to consent, and inability or unwillingness to participate regularly in the exercise program;
* unable to communicate in English or Spanish, or unlikely to fully comply with the follow-up protocol (e.g., lack of caregiver support to safely perform exercise tasks at home or complete the questionnaires).

Clarifying exclusion criteria

* Ongoing treatment: The investigators will NOT exclude those who are participating in standard of care physical therapy program (Receipt of Physical Therapy (PT), Occupational Therapy (OT), Speech Therapy (ST), Mental Health (MH), and Social Work (SW) Services). However, the investigators will document these services and will control for it. However, those who are receiving non- standard of care exercise therapy (e.g. other exercise research study) or receiving active intensive or induction therapy for cancer (e.g. undergoing active initial chemotherapy or radiotherapy).
* Others: The investigators will NOT exclude but will document common comorbidities such as pneumonia, heart failure, and chronic obstructive pulmonary disease exacerbations. Pulmonary embolism or acute coronary syndrome maybe included if there is no contraindications like severe hemodynamic instability or active angina.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Exercise dropout rate | The time frame will be from enrollment to within the first week of inpatient stay
  The investigators will evaluate feasibility of Tele-Exergame objectively by documenting the daily missed exercise session and exercise dropout within the first week of inpatient stay.

SECONDARY OUTCOMES:
Katz Activities of Daily Living Scale | The time frame will be from enrollment to 4 weeks post discharge
  The investigators will assess deconditioning and patient reported community mobility by the Katz Activities of Daily Living Scale questionnaire at baseline, within the first week of inpatient stay and at 4 weeks.

OTHER OUTCOMES:
Measuring cognition (MOCA) scale | The time frame will be from enrollment to 4 weeks post discharge
  The MOCA ( Montreal Cognitive Assessment Scale) will be used to measure cognition at baseline, within the first week of inpatient stay and at 4 weeks .

CONTACTS AND LOCATIONS:
Overall Officials: Sarvari V Yellapragada, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT04743401/ICF_000.pdf